CLINICAL TRIAL: NCT05032547
Title: Primary Care Online Emotion-regulation Treatment
Acronym: POET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Bjureberg, Med Dr, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POETF2022
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Care Online Emotion-Regulation Treatment (Experimental): The youth component in the experimental condition will include psychoeducation, addressing maladaptive beliefs about emotions and emotion regulation, and teaching adaptive emotion regulation strategies, such as mindfulness practice and acceptance of emotions and flexible cognitive reappraisal. The parent component will include psychoeducation and teaching effective responding to their children's and their own emotions.
  Interventions: Behavioral: Therapist-supported digitally delivered transdiagnostic emotion regulation treatment
- Supportive Treatment (Active Comparator): The intervention will be delivered in a blended treatment format combining asynchronous therapist-guided online modules (text/videos/audio/messaging function) with a synchronous session delivered over video-link.
  Interventions: Behavioral: Therapist-supported digitally delivered supportive treatment

INTERVENTIONS:
Behavioral: Therapist-supported digitally delivered transdiagnostic emotion regulation treatment — Please see description of experimental arm (arm one)
  Arms: Primary Care Online Emotion-Regulation Treatment
Behavioral: Therapist-supported digitally delivered supportive treatment — Please see description of active comparator arm (arm two)
  Arms: Supportive Treatment

SUMMARY:
We will evaluate a transdiagnostic digital emotion regulation treatment for youth with mental health problems.

DETAILED DESCRIPTION:
Mental health problems in youth are a global problem, causing incalculable suffering in youth and families, harming long-term prospects of youths, and are creating substantial economic costs to society. Existing treatments are not fully addressing these problems because they focus on a subset of mental health problems; they are limited in efficacy; and are not provided to most youth in need. Transdiagnostic digital treatments that address mechanisms underlying mental health problems, such as emotion regulation, have been called for to address these problems. As an initial pilot study we will include 60 participants aged 12-17 years and their parents in a randomized controlled feasibility trial comparing a 6-week Primary care Online Emotion-regulation Treatment (POET) to a 6-week active Supportive Treatment (ST). Both interventions will be delivered in blended format combining online therapist-supported treatment modules with a video-link session. The primary study aims are to examine the feasibility and acceptability of study protocol and treatment protocols. Preliminary utility of the experimental condition will be evaluated by youth-reported, parent-reported, and clinical-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with mental health problems

Exclusion Criteria:

* Acute suicidality and severe mental illness that require specialized care

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Completion of assessments | End of treatment 6 weeks after baseline
  Completion of follow-up will be defined as completing at least one clinical outcome at end of intervention.
The fraction of eligible participants who consent to inclusion and randomization | End of treatment 6 weeks after baseline
  We will determine the fraction of potential participants as the number of eligible persons compared to the number of randomized persons.
Compliance | End of treatment 6 weeks after baseline
  Compliance with the experimental intervention will be defined as completing at least three of six modules/sessions.
Child version or the Cognitive Emotion Regulation Questionnaire as explorative primary clinical outcome | Change from baseline, once every week during treatment (0-6 weeks after baseline)
  Measure of emotion regulation
Revised Child Anxiety and Depression Scale as explorative primary clinical outcome | Change from baseline, once every week during treatment (0-6 weeks after baseline)
  Measure of anxiety and depression symptoms

SECONDARY OUTCOMES:
Children's Global Assessment Scale | Change from baseline, 6 weeks after treatment starts
  Measure of global functioning
Strengths and Difficulties Questionnaire | Change from baseline, 6 weeks after treatment starts
  Measure of youth strengths and difficulties
Brief 16-item Version of the Difficulties In Emotion Regulation | Change from baseline, 6 weeks after treatment starts
  Measure of difficulties in emotion regulation
Emotion Regulation Questionnaire Child/Adolescents Version | Change from baseline, 6 weeks after treatment starts
  Measure of difficulties in cognitive reappraisal and suppression
Beliefs About Emotions Questionnaire | Change from baseline, 6 weeks after treatment starts
  Measure of beliefs about emotions
Emotion Regulation Diversity Index | Change from baseline, 6 weeks after treatment starts
  Measure of emotion regulation flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bjureberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Gustavsberg's Vårdcentral, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sjoblom K, Frankenstein K, Klintwall L, Nilbrink J, Zetterqvist M, Hesser H, Hedman-Lagerlof E, Gross JJ, Hellner C, Bellander M, Bjureberg J. Online Transdiagnostic Emotion Regulation Treatment for Adolescents With Mental Health Problems: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2514871. doi: 10.1001/jamanetworkopen.2025.14871. PMID 40498482